CLINICAL TRIAL: NCT02206152
Title: A Randomized Double Blinded Study to Examine the Use of N-Acetyl Cysteine for the Prevention and Treatment of HAAF in Patients With Type 1 Diabetes
Acronym: NAC for HAAF
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: Protocol 22498
Record Dates: First submitted 2014-05-23; First posted 2014-08-01 (Estimated); Results first posted 2020-01-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Type 1 Diabetes; Hypoglycemia Unawareness
Keywords: Diabetes; Hypoglycemia; Unawareness; HAAF
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Hypoglycemia; Unconsciousness | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Normal Saline IV infusion given during a controlled hyperinsulinemic hypoglycemic insulin clamp
  Interventions: Drug: Placebo
- Treatment with N-Acetyl Cysteine (Experimental): N-acetyl cysteine IV infusion given as a 150 mg/kg loading dose over the first hour and then follow that with a 50 mg/kg maintenance dose infused over the next 4 hours during a controlled hyperinsulinemic hypoglycemic insulin clamp
  Interventions: Drug: N-acetyl cysteine

INTERVENTIONS:
Drug: N-acetyl cysteine — N-acetyl cysteine (or saline) IV infusion given as a 150 mg/kg loading dose over the first hour and then follow that with a 50 mg/kg maintenance dose infused over the next 4 hours during a controlled hyperinsulinemic hypoglycemic insulin clamp
  Other Names: NAC
  Arms: Treatment with N-Acetyl Cysteine
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a single center, double blind randomized cross over design trial that will compare the impact of N-acetyl cysteine (200 mg) vs. saline infusion during experimental hypoglycemia on day one on the responses to experimental hypoglycemia on day two. 18 participants will be studied twice, 8 weeks apart. On each occasion they will undergo a 2 hour hypoglycemic clamp (target 50 mg/dl) in the morning and in the afternoon on day one and then again on the morning of day 2 and day 3. During the morning clamps, samples will be collected for later measurement of serum epinephrine levels, plasma and red blood cell NAC, cysteine, and glutathione concentrations and GSH/GSSG ratios (redox status), and participants will be asked to complete a hypoglycemia symptom questionnaire

DETAILED DESCRIPTION:
This study will consist of a screening visit and two 2-day intervention visits separated by approximately 8 weeks.

At the screening visit, informed consent will be obtained, a standardized form will be used to ensure subjects meet inclusion/exclusion criteria, and baseline hemoglobin A1c will be obtained. On arrival, two IVs will be placed and they will be randomized to receive NAC or saline infusion. Baseline blood samples will be drawn for glucose, epinephrine, norepinephrine, cortisol, cysteine and glutathione measurements. Subjects will then be given 25 mg IV diphenhydramine (Benadryl) followed by a 60 minute infusion of NAC (150 mg) or a similar volume of saline between 8 am and 9 am, followed by a four hour infusion of 50 mg of NAC. Thirty minutes after the start of the NAC infusion, a hyperinsulinemic (2.0 mu/kg/min) hypoglycemic (target = 50 mg/dl) clamp protocol will be started. During the morning study, blood samples will be collected every 5 minutes for monitoring of blood glucose levels and every 15 minutes for later measurement of serum epinephrine, norepinephrine, cortisol. Plasma and red blood cells samples will also be collected every 15 minutes for later measurement of NAC, cysteine, glutathione, and GSH/GSSG ratios (redox status). During the final 15 minutes of the morning clamp, subjects will be asked to quantitate their symptoms using a standardized method (13). At the completion of the morning clamp, glucose will be given to return the participant to euglycemia. 2 hours after the end of the morning clamp, a second hyperinsulinemic (2.0 mu/kg/min) hypoglycemic (target = 50 mg/dl) clamp protocol will be followed over two hours. . The afternoon clamp study will proceed as in the morning except that no serum or plasma will be collected except for the monitoring of glucose and collection of samples for subsequent measurement of NAC, cysteine, glutathione, and GSH/GSSG ratios. After the completion of the afternoon clamps, subjects will be returned to euglycemia and fed a meal. They will be discharged home.

At 7 AM the following morning they will under a single 2 hour hyperinsulinemic hypoglycemic stepped clamp (75, 65, 55,45 mg/dl targets) during which blood samples will be collected as on the morning of day 1. Symptom scores will be collected in the final 15 minutes of each step in the clamp.

At the completion of the study on day 2 of Part 1, they will be scheduled to return for Part 2 in 8 weeks. This timing is selected to ensure that female participants are studied at the same phase of the menstrual cycle. During Part 2 they will receive the treatment not provided during Part 1 in a blinded fashion. The rest of the study protocol will be the same as in Part 1.

ELIGIBILITY:
Inclusion Criteria:

* Healthy controls
* Age 18 - 65 years
* Baseline hemoglobin A1C <6.0%

Exclusion Criteria:

* History of stroke, seizures (other than those related to hypoglycemia), arrhythmias, active cardiac disease (all of which could be associated with adverse cardiac or neurological events during hypoglycemia)
* Pregnancy or plan to become pregnant during the study period
* Diagnosis of asthma (increases risk of hypersensitivity reactions to NAC)
* Use of anti-oxidants or drugs that can alter glucose metabolism
* Concomitant medical problems that may prevent the subject from successfully completing the protocol
* Unwillingness to avoid exercise during the 7 days before each part of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Seaquist, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Department of Medicine, Division of Diabetes, Endocrinology and Metabolism, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Crossover design
Groups:
- All Participants: Crossover design: All participants included in baseline data.
Period: Pre-Randomization
Arm/Group | All Participants
Started | 22
Completed | 20
Not Completed | 2
Not completed — Withdrawal by Subject | 2
Period: Placebo, Then NAC
Arm/Group | All Participants
Started | 10
Completed | 10
Not Completed | 0
Period: NAC, Then Placebo
Arm/Group | All Participants
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: This is a cross-over trial. All participants for whom baseline data was collected (20 out of 22) are pooled and reported here.
Groups:
- All Subjects: All participants at baseline
Arm/Group | All Subjects
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.7 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Difference in Epinephrine Secretion During the Morning Episodes of Hypoglycemia on Days One and Two Under the Two Treatment Conditions
Description: Epinephrine secretion during hypoglycemia is assessed by collecting blood samples for measurement of epinephrine concentrations at baseline and every 15 minutes during the period of hypoglycemia (starting at point where blood glucose is first < 55 mg/dl) in the clamp studies done in the mornings of days 1 and 2 of both parts 1 and 2. .
Time Frame: 8-10 weeks
Measure: Mean (Standard Deviation); unit: ug/ml
Groups:
- Placebo: Normal Saline IV infusion given during a controlled hyperinsulinemic hypoglycemic insulin clamp
  Placebo
Arm/Group | Placebo | Treatment With N-Acetyl Cysteine
Number analyzed (Participants) | 20 | 20
ug/ml | 622.8 (334.1) | 867 (675.9)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Placebo | Treatment With N-Acetyl Cysteine
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 9/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=20) | Treatment With N-Acetyl Cysteine (N=20)
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 7
Nausea (Gastrointestinal disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-10-12): https://cdn.clinicaltrials.gov/large-docs/52/NCT02206152/Prot_SAP_000.pdf
  • Informed Consent Form (2017-06-15): https://cdn.clinicaltrials.gov/large-docs/52/NCT02206152/ICF_001.pdf